CLINICAL TRIAL: NCT06565806
Title: French National Cohort of Patients With Rifampicin-Resistant Tuberculosis
Acronym: CONTRol-TB
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240748
Record Dates: First submitted 2024-08-12; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Rifampicin-resistant Tuberculosis
Keywords: Tuberculosis; Rifampicin-resistant
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Retrospective cohort 2006-2019
- Retrospective cohort of the CNR national register of Mycobacteria from 2020 to end of May 2024
- Prospective cohort of the CNR national register of Mycobacteria from June 2024 to the end of 2029

SUMMARY:
A major obstacle in the fight against multidrug-resistant tuberculosis is its treatment. In 2021, only 60% of patients with MDR/RR tuberculosis who received treatment globally were successfully cured, while 12% succumbed to the disease and 10% experienced treatment failure.

In France, a recent study by the National Reference Centre for Mycobacteria showed that while MDR/RR tuberculosis patients treated between 2006 and 2019 in the major reference centres in the Paris region achieved a favourable outcome in 68% of cases, 30% were lost. The main aim of this study is to enhance our understanding of the outcomes for patients suffering from tuberculosis due to rifampin-resistant bacilli, as well as the factors influencing these outcomes. Additionally, it aims to decrease the duration required to relay information to health authorities regarding the status of multidrug resistance and the outcomes of patients in France.

A national longitudinal cohort will be develop to study multidrug-resistant tuberculosis in France. The cohort includes a historical retrospective part from 2006-2019 and a prospective part from 2020, with planned inclusions until 2029. The restrospective cohort includes 298 patients from 2006-2019 and 178 patients from the CNR mycobacteria national registry until 2024. As for the prospective cohort arm, a projected total of roughly 300 patients will be included over the period from 2020 to 2029. Non-identifying clinical data will be derived exclusively from patients medical records at three expert centres in the Paris region for the restrospective cohort and throughout France (national register) for the prospective cohorte. For the retropective cohorte each centers will transcribe pseudonymised clinical data into secure Excel files, while the prospective cohort will enter non-identifying data directly into the national register using a secure platform overseen by the CNR of Mycobactéria.

Registry data will be extracted directly from the registry and merged with the retrospective database every 12 months by the coordinating investigator. Statistical analyses will include descriptive analyses of continuous and categorical variables, comparisons between subgroups using appropriate tests (Student's t, Mann-Whitney, Chi Square, Fisher), and logistic regressions to identify variables associated with treatment outcomes. P value < 0.05 will be considered statistically significant

DETAILED DESCRIPTION:
Tuberculosis (TB) is a major global health problem. Over the past decade, Mycobacterium tuberculosis has killed more people worldwide than any other infectious pathogen, and drug-resistant TB accounts for a third of deaths linked to antimicrobial resistance (AMR). A major obstacle in the fight against multidrug-resistant tuberculosis is its treatment. In 2021, only 60% of patients with MDR/RR tuberculosis who received treatment globally were successfully cured, while 12% succumbed to the disease and 10% experienced treatment failure. In France, a recent study by the National Reference Centre for Mycobacteria showed that while MDR/RR tuberculosis patients treated between 2006 and 2019 in the major reference centres in the Paris region achieved a favourable outcome in 68% of cases, 30% were lost.

In a context of low incidence and loss of expertise in the management of MDR/RR tuberculosis in Western Europe and France, the creation of a national retrospective and prospective cohort will make it possible to measure the treatment outcomes of these patients, a vital indicator for assessing the quality of care.The main aim of this study is to enhance our understanding of the outcomes for patients suffering from tuberculosis due to rifampin-resistant bacilli, as well as the factors influencing these outcomes. Additionally, it aims to decrease the duration required to relay information to health authorities regarding the status of multidrug resistance and the outcomes of patients in France

This is a national longitudinal cohort which includes a historical retrospective part (2006-2019) and a prospective part developed with the setting up of the CNR national register of Mycobacteria (from 2020, planned inclusions until 2029). The population in the restrospective cohort includes 298 patients in the period 2006-2019 and 178 included in the national registry of the CNR mycobacteria national registry till end of May 2024. As for the prospective cohort arm, a projected total of roughly 300 patients will be incorporated over the period from 2020 to 2029. Non-identifying clinical data for the restrospective cohorte will be exclusively derived from the medical records of patients, in the investigating departments of the 3 expert centres for multidrug-resistant tuberculosis in the Paris region (Hôpitaux de la Pitié-Salpêtrière, Bichat and Bligny). Each centre will transcribe its own pseudonymised clinical data into a secure Excel file, which will then be transmitted via Dispose AP-HP to the coordinating investigator, and stored on a secure computer at the CNR of Mycobactéria.

For the prospective cohort the non-identifying clinical data will be entered directly by patient referral departments into the CNR des Mycobactéries national register, on a secure platform developed specifically for the register and managed by the CNR of Mycobactéria. Any department in charge of patients with multidrug-resistant tuberculosis in France will be able to take part in prospective inclusion in the register.

Registry data will be extracted directly from the registry and merged with the retrospective database every 12 months by the coordinating investigator. Statistical analyses will include descriptive analyses of continuous and categorical variables, comparisons between subgroups using appropriate tests (Student's t, Mann-Whitney, Chi Square, Fisher), and logistic regressions to identify variables associated with treatment outcomes. P value < 0.05 will be considered statistically significant

ELIGIBILITY:
Inclusion Criteria:

Patient treated for MDR/RR tuberculosis

* In the major reference centres in the Paris region (CHU Pitié-Salpêtrière and Bichat [Paris], CH Bligny [Briis-sous-Forges]) for the retrospective part;
* Throughout France (national register) for the prospective part.

Exclusion Criteria:

* None

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patient treated for MDR/RR tuberculosis in the major reference centres in the Paris region and throughout France (national register).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2029-08-01 (Estimated); Study Completion 2032-09-01 (Estimated)

PRIMARY OUTCOMES:
Outcome of tuberculosis treatment (WHO 2021 outcome definitons) | Through out study time period (Till 2029)

SECONDARY OUTCOMES:
Prognostic factors in the evolution of tuberculosis | Through out study time period (Till 2029)

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request The procedures carried out with the French data privacy authority (CNIL) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.